CLINICAL TRIAL: NCT05228535
Title: Early Fortification of Human Milk for Very Low Birth Weight Infants and Effects on Growth Velocity
Brief Title: Human Milk in Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1813934-2
Record Dates: First submitted 2022-01-14; First posted 2022-02-08 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: 2 groups. 1 group will be controlled, following standard NICU feeding protocol. 1 group will be intervention, receiving early introduction of human milk fortifier to enteral feeds.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Continue current NICU feeding protocol, introducing human milk fortifier at 8 days
- Intervention (Experimental): Introducing human milk fortifier at 1 day
  Interventions: Dietary Supplement: Human milk fortifier

INTERVENTIONS:
Dietary Supplement: Human milk fortifier — Human milk fortifier added to human breast milk at day 1 vs day 8 of feeds
  Arms: Intervention

SUMMARY:
Current NICU protocol introduces human milk fortifier at 8 days of feeding. This study will introduce human milk fortifier at day 1. The primary outcome is the effect on growth velocity at 28 days and 36 weeks post menstrual age.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight 1000-1500 grams
* Admitted to NICU within 24 hours of life
* Maternal intent to use human milk

Exclusion Criteria:

* Congenital anomalies
* Feeds not started within the first 96 hours of life
* Intrauterine growth restriction

Max Age: 4 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Growth velocity | at 28 days of life
  weight gain in grams/kg/day

SECONDARY OUTCOMES:
Growth velocity | at 36 weeks post menstrual age
  weight gain in grams/kg/day

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Georgia, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wynter Z, Gorham JA, Thompson AB, Mundy C, Waller JL, Stansfield BK. Immediate fortification of human milk with a bovine milk-derived human milk fortifier in very low birth weight infants: a randomized clinical trial. J Perinatol. 2024 Nov;44(11):1591-1596. doi: 10.1038/s41372-024-01998-0. Epub 2024 May 9. PMID 38724605

DOCUMENTS (2):
  • Study Protocol (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT05228535/Prot_000.pdf
  • Informed Consent Form (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT05228535/ICF_001.pdf